CLINICAL TRIAL: NCT04232761
Title: Safety and Effectiveness of Xofigo® (Radium-223 Dichloride) in Routine Clinical Practice Settings in Taiwan
Brief Title: Study to Gather Information on the Safety and How Radium-223 Dichloride, an Alpha Particle-emitting Radioactive Agent, Works Under Routine Clinical Practice in Taiwan in Patients With Castration-resistant Prostate Cancer (CRPC) Which Has Spread to the Bone
Acronym: RAPIT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21124
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Bone metastases; Radium-223 dichloride
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRPC patients: Patients with castration-resistant prostate cancer (CRPC) and symptomatic bone metastases who are treated with radium-223 dichloride in routine clinical practice in Taiwan
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Drug administration as determined by treating physician

SUMMARY:
In this observational study researchers want to gather more information about safety and survival in patients suffering from castration-resistant prostate cancer (CRPC) which has spread to the bone and were treated with radium-223 in routine clinical practice in Taiwan. Radium-223 (Ra-223) is an alpha particle-emitting radioactive agent approved for the treatment of men with metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
The primary objective of the study is to describe the safety profile of radium-223 dichloride in patients having castration-resistent prostate cancer with symptomatic bone metastases and who are treated in routine clinical practice in Taiwan.

The secondary objective is to assess the effectiveness of radium-223 dichloride in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed castration-resistant adenocarcinoma of the prostate with bone metastases
* Treatment decision for Radium-223 according to local label needs to be made independent from and before patient enrollment in the study by the investigator
* No contra-indications according to the local marketing authorization

Exclusion Criteria:

* Previously treated with Radium-223 for any reason
* Currently treated in clinical trials including other Radium-223 studies or planned participation in an investigational program with interventions outside of routine clinical practice during the study period

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients in routine clinical practice from Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 7 months
Incidence of drug-related TEAEs | Up to 7 months
Descriptive analysis of long-term safety information during the extended follow-up period | Up to 2 years
  This safety information may include e.g. hematological adverse events, bone fractures or osteoporosis.

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
Time to the first symptomatic skeletal event (SSE) | Up to 2 years
Proportion of patients with total ALP (tALP) response | Up to 2 years
  ALP - Alkaline Phosphatase tALP - Total Alkaline Phosphatase
Proportion of patients with PSA response | Up to 2 years
  PSA - Prostate Specific Antigen
Change in pain status | Up to 2 years
  Pain status is assessed through analgesic utility that is calculated by WHO analgesic scores (0 - none, 1 - non-opioid, 2 - opioid for mild to moderate pain, 3 - opioid for moderate to severe pain)
Change in ECOG-PS | Up to 2 years
  The Cooperative Oncology Group-Performance Status (ECOG-PS) score ranks the performance status from 0 (perfect health) to 5 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Taiwan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.